CLINICAL TRIAL: NCT00675376
Title: Lung Transplant for COPD: Outcomes/Technology
Brief Title: Evaluating Quality of Life for Patients With Chronic Obstructive Pulmonary Disease Who Are Undergoing Lung Transplantation
Status: Terminated | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 564; R01HL083067 (NIH)
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Lung Transplantation
Keywords: COPD; Lung Transplant; Quality of Life; End Stage Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Most people undergoing lung transplantation have chronic obstructive pulmonary disease (COPD), a disease in which the lung airways are partly damaged and obstructed, making it difficult to breathe. This study will enroll people with COPD who are undergoing a lung transplant to examine how their quality of life changes after the transplant procedure.

DETAILED DESCRIPTION:
Lung transplantation is one treatment option for people with end-stage lung disease. The majority of people undergoing a lung transplant have COPD, and while transplantation can potentially improve survival and quality of life, it may also carry substantial risks, including surgical complications, infections, and pneumonia. The impact of lung transplantation on survival and quality of life has not been extensively studied. In the United States, the United Network for Organ Sharing (UNOS) is the organization that allocates donor lungs to lung recipients. Before 2005, the length of time that a candidate had been on the transplant waiting list was the major determining factor for receiving a donor lung. In mid 2005, the UNOS system changed and began prioritizing candidates on the basis of risk of death prior to lung transplantation and the probability of death within the first year after transplantation. The purpose of this study is to evaluate quality of life factors for lung transplant patients with COPD, both before and after the lung transplant procedure. In addition, quality of life of patients in the new UNOS allocation system will be compared with that of patients in the old UNOS allocation system.

This study will enroll all COPD patients undergoing an evaluation for lung transplantation at the Washington University Medical Center and Barnes-Jewish Hospital in St. Louis, Missouri. Participants will attend study visits at the time of the transplant evaluation and again just prior to listing in the UNOS system. After the transplant, participants will attend study visits at Months 3 and 6 and then once a year for 5 years. During each study visit, participants will complete a computerized interview and health-related questionnaires that will assess quality of life factors, including social life, work life, and home life. Study researchers will also review participants' medical records to collect information on lung function and blood test results.

ELIGIBILITY:
Inclusion Criteria:

* Referred to the adult lung transplant program
* Undergoing evaluation for lung transplantation
* Very severe COPD (Global Initiative for Chronic Obstructive Lung Disease [GOLD] class IV) that is predominantly due to emphysema
* Able to read English
* Able to adequately see a computer screen

Exclusion Criteria:

* Diagnosis other than COPD
* Inability to read English

Ages: 21 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study participants will undergo evaluation in the lung transplant clinic at Washington University Medical Center and Barnes-Jewish Hospital. They must have the diagnosis of COPD predominantly due to emphysema.
Sampling Method: Non-Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2006-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Assessment of the effectiveness of lung transplantation in patients with COPD in the new donor lung allocation system | Measured throughout the study

SECONDARY OUTCOMES:
Comparison of the effects of lung transplantation on the quality of life of patients with COPD in the new donor lung allocation system versus the old donor lung allocation system | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Roger D. Yusen, MD, MPH, Principal Investigator — Washington University School of Medicine, St. Louis
Locations (1):
- Washington University School of Medicine and Barnes-Jewish Hospital, St Louis, Missouri, United States